CLINICAL TRIAL: NCT04665557
Title: Evaluating "Dove Confident Me Indonesia"; A School-Based Single Session Intervention to Improve Body Image and Wellbeing Among Indonesian Adolescents
Brief Title: Evaluating Dove Confident Me Single Session in Indonesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the West of England (Other)
Collaborators: Indonesia University (Other); University of Hawaii (Other); UNICEF (Other); Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DSEP_UNICEF_INDO; HAS-HSS-18-098 (Other: University of the West of England, PASS reference)
Record Dates: First submitted 2020-09-29; First posted 2020-12-11 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Body Image

STUDY DESIGN:
Intervention Model Description: Two-arm parallel clustered randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Masking not possible for participants within design, but outcome assessors will not know what condition participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dove Confident Me Indonesia - Single Session (Experimental): Dove Confident Me Indonesia Single Session is school-based, body image curriculum.
  Interventions: Behavioral: Dove Confident Me Indonesia Single Session
- Lessons As Usual Control (No Intervention): School lessons as usual.

INTERVENTIONS:
Behavioral: Dove Confident Me Indonesia Single Session — Dove Confident Me Indonesia Single Session is an adaptation of Dove Confident Me Global Single Session, designed to be facilitated by schoolteachers or school counsellors. Dove Confident Me Indonesia includes four interactive activities (to be delivered in a single 90-minute session) as well as a homework challenge and commitment pledge. The programme incorporates three primary techniques to improve Indonesian adolescents' body confidence and self-esteem: (1) psychoeducation, (2) media literacy, and (3) cognitive dissonance as well as two secondary techniques: (4) self-affirmation and (5) cognitive reframing. As the curriculum was adapted to be delivered in Indonesian schools with limited resources, videos or PowerPoint presentations are not included. Instead, a detailed teacher guide and student worksheets are provided.
  Due to COVID-19, the intervention will be delivered online via video conferencing platform.
  Arms: Dove Confident Me Indonesia - Single Session

SUMMARY:
Negative body image is an important public health concern for young people due to its prevalence and detrimental impact on young people's health, education, and social life. Encouragingly, a number of interventions have been designed to improve adolescent body image in school settings, with promising results. However, the vast majority of studies testing these interventions are conducted in high-income, English speaking countries, despite increasingly recognition that negative body image is a global concern. As such, it is important to develop and disseminate interventions to foster positive body image among adolescents in low-to-middle income countries, too.

Research indicates high prevalence rates of negative body image among adolescents in many Asian countries. Indonesia - the focus of the present research - is an emerging middle-income country in South East Asia. A recent U-Report Poll (UNICEF, 2020) found almost 80% of the young people surveyed wanted to change something about their appearance, suggesting a degree of body dissatisfaction and approximately 50% stopped themselves from doing something that was important to them because of appearance concerns. Moreover, according to the same poll, over 90% of Indonesian adolescents surveyed reported to wanting to learn ways to improve their body image in school or online.

To date, no body image interventions have been adapted and trialled in Indonesia. Therefore, this project aims to evaluate the effectiveness as well as the acceptability and feasibility of a specially adapted version of Dove Confident Me Single Session among Indonesian adolescents that will be integrated into UNICEF's Life Skills Education curriculum. Notably, the session has been designed to be feasible to deliver in low-resource schools (e.g., that do not access to the internet or facilities to show videos or PowerPoint slides).

To assess the acceptability, feasibility, and effectiveness of the intervention, the study will compare the body image and well-being of students who take part in the programme to students who do not take part in any programme (classes as usual). Investigators will also gather in-depth feedback from students, and teachers via focus groups and surveys, in order to inform future improvement of the programme for wider implementation.

To undertake this project, the investigators will recruit students and teachers from approximately 10 state junior secondary schools in Indonesia via a local research agency. Students will complete questionnaire assessments of body image and well-being before and after programme period, and again 8 weeks later to assess longer-term benefits.

COVID response: In light of the ongoing pandemic, some research activities will take place online. Decisions on delivery format (online / in-person / hybrid) were made on the basis of continued risk assessments and considerations of local government guidelines.

DETAILED DESCRIPTION:
Detailed COVID Response Description. Though the intervention was specifically designed to be delivered in person and avoided the use of technology to make it accessible to as many Indonesian adolescents as possible, circumstances with COVID-19 have meant that aspects of trial need to be conducted online to minimise undue harm and the spread of infection. Decisions on delivery format were based on regular risk assessments and considerations of local government guidelines. Accordingly, the internal pilot was conducted entirely online as most schools were exclusively offering remote learning and the risk in the area was high. In contrast, shortly following the commencement of the main trial, schools in Surabaya returned to 100% in person teaching (January 2022). Consequently, some research activities, including the lesson, took place in school while sticking to health and safety measures (e.g., social distancing, wearing masks, etc.).

Teacher training will include self-directed learning via UNICEF's teacher training e-module for Life Skills Curriculum which includes the intervention of focus on body image. Teachers will then attend two online training sessions with a member of the research team who is trained in delivering the intervention. These sessions will run through background knowledge about body image, propose how we expect the lesson to look, give the opportunity for teachers to ask questions, and explore common questions/statements from students.

Schools will be recruited for the study via email correspondence from the research agency in Indonesia and information sheets will be sent out to parents/guardians. Parents/guardians will provide informed consent to the school. Students will provide informed consent to the school and during the baseline assessment. Students will complete the surveys across three time points via Qualtrics on personal devices at home or at school. The acceptability focus groups with teachers and students from the intervention condition will take place via a video conferencing platform such as Zoom. The intervention will be delivered online via video conferencing platform.

To ensure this method of the trial is feasible, we need to ensure students have access to a device (laptop or iPad), have a stable internet connection and are familiar with video conferencing platforms for learning. To meet these demands, we will recruit in higher SES areas.

Further, given that we did not initially plan to conduct any aspects of the trial online, we ran an internal acceptability pilot. That is, we tested the feasibility and acceptability of key study elements - i.e., administering the surveys online across three timepoints and delivering the intervention online with two classes. Additionally, we conducted small focus groups with students to access their feedback on the intervention. If the data quality from the pilot is poor and the engagement in the lesson is low, we will suspend the trial until schools resume face to face learning and the COVID-19 risk is much lower (e.g., when there is widespread uptake of the vaccine).

ELIGIBILITY:
Inclusion Criteria:

* All participating schools must be state junior secondary schools.
* Students in grade 7 through 9 are eligible.
* Students must speak Bahasa Indonesia and must have moderate-high literacy. levels in Bahasa Indonesia - i.e., need to be able to read on their own.
* Students must have access to a device with online access (e.g., laptop or iPad).

Exclusion Criteria:

* Non-Bahasa Indonesia speaking students.
* Religious or private schools.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1926 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change in body esteem | Baseline; post intervention (1 week after the intervention) and follow-up (8 weeks after the intervention).
  Body esteem will be assessed using the weight and appearance evaluation subscales of the Body Esteem Scale for Adolescents & Adults (BESAA, Mendelson, Mendelson & White, 2001). Responses to the 18 items are on a 5-point Likert-type scale. Once the appropriate items are reverse coded, scores will be averaged with higher scores indicating higher body esteem.

SECONDARY OUTCOMES:
Change in internalisation of societal appearance ideals | Baseline; post intervention (1 week after the intervention) and follow-up (8 weeks after the intervention).
  Internalisation of societal appearance ideals will be assessed using the general subscale of the Sociocultural Attitudes Towards Appearance Questionnaire-3 (SATAQ-3; Thompson, Van Den Berg, Roehrig, Guarda, & Heinberg, 2004). Scores will be averaged with higher scores indicating higher internalisation. Mean score range = 1-5.
Change in mood | Baseline; post intervention (1 week after the intervention) and follow-up (8 weeks after the intervention).
  Positive and negative affect will be measured using the Positive and Negative Affect Schedule (Crawford & Henry, 2004). Scores on each subscale will be averaged; with higher scores indicating greater negative affect and positive affect respectively. Mean score range for each subscale = 1-5.
Change in tendency to engage in appearance comparisons | Baseline; post intervention (1 week after the intervention) and follow-up (8 weeks after the intervention).
  Two purpose-built items will assess participants' tendency to engage in appearance comparisons. Responses to both items will be on a 5-point Likert-type scale (1=Never to 5=Often). Scores will be averaged with higher scores indicating a greater tendency to engage in appearance comparisons.
Skin shade satisfaction | Baseline; post intervention (1 week after the intervention) and follow-up (8 weeks after the intervention)
  Three purpose-built items will assess participants' satisfaction with their skin shade (i.e., the precise colour of their skin). Responses to the initial two items will be on a 5-point Likert-type scale.
  'How dissatisfied or satisfied you are with the colour of your skin?' is rated from 1=very dissatisfied to 5 = very satisfied. 'Which of the following statements do you agree with the most' - 1 = I would like my skin colour to be lighter, 2 = I would like my skin colour to stay the same and 3 = I would like my skin colour to be darker.
  The final skin shade satisfaction item will use a visual representation of skin colours (1=darkest skin shade to 9=lightest skin shade). Participants will be asked which skin shade is most alike to their current skin colour, and then which skin shade is closest to their 'ideal' skin colour.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Craddock, PhD, Principal Investigator — Centre for Appearance Research, UWE
Locations (1):
- Centre for Appearance Research, UWE, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This needs to be a shared decision based on a memorandum of understanding between the University of Indonesia and the University of the West of England. This is not yet finalised.

REFERENCES:
- [Derived] Craddock N, Garbett KM, Haywood S, Nasution K, White P, Saraswati LA, Rizkiah C, Medise BE, Diedrichs PC. 'Dove Confident Me Indonesia: Single Session': study protocol for a randomised controlled trial to evaluate a school-based body image intervention among Indonesian adolescents. BMC Public Health. 2021 Nov 16;21(1):2102. doi: 10.1186/s12889-021-11770-0. PMID 34784916